CLINICAL TRIAL: NCT00015873
Title: International Collaborative Treatment Protocol for Infants Under One Year With Acute Lymphoblastic Leukemia
Brief Title: Comparison of Different Combination Chemotherapy Regimens in Treating Infants With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dutch Childhood Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068529; ICU-INTERFANT99; UKCCSG-LK-1999-05; EU-20063; EU-20588
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Asparaginase; Cytarabine; Mercaptopurine; Methotrexate; Prednisolone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A no VIMARAM (No Intervention): No VIMARAM preceding maintenance treatment
- B - VIMARAM (Experimental): VCR i.v. 1.5 mg/m2/d - 4 days 6-MP p.o. 25 mg/m2/d - 15 days HD-MTX p.i.(24hr) 5 g/m2 - 2 days MTX + pred I.T. (age adapted) - 2 days HD-Ara-C p.i (3hr) 3 g/m2/12 hrs -8 days L-ASP p.i. (1hr) 5.000 U/m2 - 2 days
  Interventions: Drug: asparaginase; Drug: cytarabine; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisolone; Drug: vincristine sulfate

INTERVENTIONS:
Drug: asparaginase
  Arms: B - VIMARAM
Drug: cytarabine
  Arms: B - VIMARAM
Drug: mercaptopurine
  Arms: B - VIMARAM
Drug: methotrexate
  Arms: B - VIMARAM
Drug: prednisolone
  Arms: B - VIMARAM
Drug: vincristine sulfate
  Arms: B - VIMARAM

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is most effective for treating infants with acute lymphoblastic leukemia.

PURPOSE: Randomized phase III trial to compare the effectiveness of different combination chemotherapy regimens in treating infants who have newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the outcome of induction chemotherapy followed by consolidation and reinduction chemotherapy with or without late intensification chemotherapy followed by a maintenance regimen or allogeneic bone marrow transplantation in infants with newly diagnosed acute lymphoblastic leukemia.
* Determine the value of a late intensification course between reinduction and maintenance therapy in these patients.
* Determine the prognostic value of age, immunophenotype, WBC, day 15 bone marrow status, and MLL gene rearrangement in patients treated with these regimens.

OUTLINE: This is a partially randomized, multicenter study. Patients are stratified according to risk (high vs standard).

Patients receive induction therapy comprising prednisone orally or IV three times a day on days 1-7; dexamethasone orally or IV three times a day on days 8-35; vincristine IV on days 8, 16, 22, and 30; cytarabine IV over 30 minutes on days 8-21; daunorubicin IV over 60 minutes on days 8 and 9; asparaginase IV over 1 hour or intramuscularly (IM) on days 15, 18, 22, 25, 29, and 33; methotrexate intrathecally (IT) on days 1 and 29; and cytarabine IT on day 15. Patients receive prednisolone IT in combination with any dose of intrathecal chemotherapy. Patients with CNS involvement receive additional doses of methotrexate IT on days 8 and 22 and then weekly after day 29 until there is no evidence of CNS leukemia.

After achieving complete remission, patients receive MARAM chemotherapy comprising oral mercaptopurine daily on days 1-14; methotrexate IV over 24 hours on days 1 and 8; leucovorin calcium orally or IV 36, 42, and 48 hours after beginning each dose of oral methotrexate; methotrexate IT on days 2 and 9; cytarabine IV over 3 hours twice daily on days 15, 16, 22, and 23; and asparaginase IV over 1 hour or IM on days 16 and 23. Patients receive prednisolone IT in combination with any dose of intrathecal methotrexate.

At least 2 weeks after the completion of MARAM chemotherapy, patients receive OCTADD chemotherapy comprising oral dexamethasone three times a day on days 1-21; oral thioguanine daily on days 1-28 and 36-49; vincristine IV on days 2, 8, 16, and 22; daunorubicin IV over 60 minutes on days 1, 8, 15, and 22; cytarabine IV on days 2-5, 9-12, 16-19, 23-26, 37-40, and 45-48; cytarabine IT on days 1 and 15; and cyclophosphamide IV over 1 hour on days 36 and 49. Patients receive prednisolone IT in combination with any dose of intrathecal methotrexate.

Patients are randomized to one of two treatment arms for late intensification therapy.

* Arm I: Beginning at least 1 week after the completion of OCTADD chemotherapy, patients receive VIMARAM chemotherapy comprising vincristine IV on days 1, 8, 15, and 22; oral mercaptopurine daily on days 1-14; methotrexate IV over 24 hours on days 1 and 8; leucovorin calcium orally or IV 36, 42, and 48 hours after the beginning of each dose of oral methotrexate; methotrexate IT on days 2 and 9; cytarabine IV over 3 hours twice daily on days 15, 16, 22, and 23; and asparaginase IV over 1 hour or IM on days 16 and 23. Patients receive prednisolone IT in combination with any dose of intrathecal methotrexate. Patients then receive the appropriate maintenance therapy.
* Arm II: Patients do not receive VIMARAM chemotherapy but receive appropriate maintenance therapy.

At least 2 weeks after the completion of the last course of chemotherapy, patients receive maintenance therapy. Patients with a good response to initial therapy with prednisone receive maintenance therapy comprising oral dexamethasone three times daily on weeks 1 and 2; vincristine IV on day 2 of weeks 1 and 2; oral mercaptopurine daily on weeks 1-14; and oral methotrexate once weekly on weeks 1-14.

Patients with a poor response to initial therapy with prednisone receive maintenance therapy comprising oral mercaptopurine daily for weeks 1-14; oral methotrexate once weekly for weeks 1-14; oral dexamethasone three times daily for weeks 1 and 2; vincristine IV on day 2 of weeks 1 and 2; etoposide IV over 2 hours once weekly on weeks 8 and 9; and cytarabine IV over 1 hour once weekly on weeks 8 and 9.

Treatment repeats in both maintenance therapy regimens every 14 weeks for a total of 3 courses. Patients also receive methotrexate IT on day 1 of the first and third course of therapy and cytarabine IT on day 1 of the second course of therapy. Patients receive prednisolone IT in combination with any dose of intrathecal chemotherapy.

Beginning after the completion of maintenance therapy, all patients receive continuing maintenance therapy comprising oral mercaptopurine daily and oral methotrexate once a week. Treatment continues until 104 weeks after initial diagnosis.

Patients with a poor response to initial therapy with prednisone may receive allogeneic bone marrow transplantation if a donor is available. The patient undergoes transplantation immediately after OCTADD chemotherapy rather than being randomized and receiving maintenance therapy. These patients receive conditioning regimen comprising oral busulfan four times a day on days -8 to -5, etoposide IV over 4 hours on day -4, methotrexate IT on day -3, and cyclophosphamide IV over 1 hour on days -3 and -2. Allogenic bone marrow is transplanted on day 0. Patients then receive cyclosporine orally or IV on days 1-180 as graft-versus-host disease prophylaxis.

Patients are followed annually.

PROJECTED ACCRUAL: A total of 350 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL)

  * Newly diagnosed
  * Morphological verification by cytochemistry and immunophenotyping
* CNS or testicular leukemia at diagnosis allowed
* Trisomy 21 allowed

PATIENT CHARACTERISTICS:

Age:

* 365 days or less

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for leukemia

Endocrine therapy:

* At least 4 weeks since prior systemic corticosteroids
* Prior inhaled steroids allowed

Radiotherapy:

* No prior radiotherapy for leukemia

Surgery:

* Not specified

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 1999-05; Primary Completion 2006-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Event-free survival at 3-4 years after diagnosis | 4 years after diagnosis
  Event-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Rob Pieters, MD, MSC, PhD, Study Chair — Erasmus MC-Sophia Children's Hospital
Locations (33):
- United States (2):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- St. Anna Children's Hospital, Vienna, Austria
- Hopital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium
- University Hospital Motol, Prague, Czechia
- Hopital Saint-Louis, Paris, France
- Germany (2):
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- Italy (2):
  - Nuovo Ospedale San Gerardo at University of Milano-Bicocca, Monza
  - Ospedale San Gerardo, Monza
- Erasmus MC - Sophia Children's Hospital, Rotterdam, Netherlands
- Ostra Sjukhuset, Gothenburg, Sweden
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton University Hospital NHS Trust, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Result] Hempel G, Relling MV, de Rossi G, Stary J, De Lorenzo P, Valsecchi MG, Barisone E, Boos J, Pieters R. Pharmacokinetics of daunorubicin and daunorubicinol in infants with leukemia treated in the interfant 99 protocol. Pediatr Blood Cancer. 2010 Mar;54(3):355-60. doi: 10.1002/pbc.22266. PMID 19731319
- [Result] Mann G, Attarbaschi A, Schrappe M, De Lorenzo P, Peters C, Hann I, De Rossi G, Felice M, Lausen B, Leblanc T, Szczepanski T, Ferster A, Janka-Schaub G, Rubnitz J, Silverman LB, Stary J, Campbell M, Li CK, Suppiah R, Biondi A, Vora A, Valsecchi MG, Pieters R; Interfant-99 Study Group. Improved outcome with hematopoietic stem cell transplantation in a poor prognostic subgroup of infants with mixed-lineage-leukemia (MLL)-rearranged acute lymphoblastic leukemia: results from the Interfant-99 Study. Blood. 2010 Oct 14;116(15):2644-50. doi: 10.1182/blood-2010-03-273532. Epub 2010 Jun 30. PMID 20592248
- [Result] Lonnerholm G, Valsecchi MG, De Lorenzo P, Schrappe M, Hovi L, Campbell M, Mann G, Janka-Schaub G, Li CK, Stary J, Hann I, Pieters R; Interfant-99 study group. Pharmacokinetics of high-dose methotrexate in infants treated for acute lymphoblastic leukemia. Pediatr Blood Cancer. 2009 May;52(5):596-601. doi: 10.1002/pbc.21925. PMID 19132729
- [Result] van der Linden MH, Valsecchi MG, De Lorenzo P, Moricke A, Janka G, Leblanc TM, Felice M, Biondi A, Campbell M, Hann I, Rubnitz JE, Stary J, Szczepanski T, Vora A, Ferster A, Hovi L, Silverman LB, Pieters R. Outcome of congenital acute lymphoblastic leukemia treated on the Interfant-99 protocol. Blood. 2009 Oct 29;114(18):3764-8. doi: 10.1182/blood-2009-02-204214. Epub 2009 Aug 5. PMID 19657114
- [Result] Van der Velden VH, Corral L, Valsecchi MG, Jansen MW, De Lorenzo P, Cazzaniga G, Panzer-Grumayer ER, Schrappe M, Schrauder A, Meyer C, Marschalek R, Nigro LL, Metzler M, Basso G, Mann G, Den Boer ML, Biondi A, Pieters R, Van Dongen JJ; Interfant-99 Study Group. Prognostic significance of minimal residual disease in infants with acute lymphoblastic leukemia treated within the Interfant-99 protocol. Leukemia. 2009 Jun;23(6):1073-9. doi: 10.1038/leu.2009.17. Epub 2009 Feb 12. PMID 19212338
- [Result] Pieters R, Schrappe M, De Lorenzo P, Hann I, De Rossi G, Felice M, Hovi L, LeBlanc T, Szczepanski T, Ferster A, Janka G, Rubnitz J, Silverman L, Stary J, Campbell M, Li CK, Mann G, Suppiah R, Biondi A, Vora A, Valsecchi MG. A treatment protocol for infants younger than 1 year with acute lymphoblastic leukaemia (Interfant-99): an observational study and a multicentre randomised trial. Lancet. 2007 Jul 21;370(9583):240-250. doi: 10.1016/S0140-6736(07)61126-X. PMID 17658395
- [Result] Pieters R, Schrappe M, de Lorenzo P, et al.: Outcome of infants less than one year of age with acute lymphoblastic leukemia treated with the Interfant-99 protocol. [Abstract] Blood 108 (11): A-145, 2006.